CLINICAL TRIAL: NCT05599165
Title: Speech Perception Enhancement Using Novel Signal Processing in Bimodal Hearing
Brief Title: Speech Perception in Bimodal Hearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: Baylor Scott and White Health (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1001262; 1R15DC019240-01A1 (NIH)
Record Dates: First submitted 2022-10-12; First posted 2022-10-31 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: A single group of bimodal cochlear implant users will be tested with three different signal processing for consonant enhancement in noise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- signal processing on consonant recognition (Experimental): The effects of the three processing schemes on consonant enhancement will be measured.
  The results will be compared with two signal processing schemes: target-cue signal processing, and combined target and conflict-cue signal processing.
  Interventions: Other: signal processing on consonant recognition

INTERVENTIONS:
Other: signal processing on consonant recognition — Consonant recognition will be measured in noise without any signal processing.

SUMMARY:
The protocol has two aims; Aim 1 involves two experiments and Aim 2 involves three experiments. Under Aim 1, the investigator will identify that the frequency and time ranges of consonants produce consonant enhancement (i.e., "target frequency range" and "target time range", respectively), and that the frequency and time ranges of consonants cause consonant confusions (i.e., "conflicting frequency range" and "conflicting time range", respectively). Aim 2 tests the effects of the frequency and time ranges, identified through Aim 1 on consonant recognition with each of the four signal processing conditions: no signal processing (i.e., control condition), the target frequency and time ranges intensified alone, the conflicting frequency and time ranges suppressed alone, and both target range intensification and conflicting range suppression.

DETAILED DESCRIPTION:
Speech perception for those who use cochlear implants (CIs) in combination with hearing aids (HAs) in opposite ears (i.e., bimodal hearing) varies greatly. This variability depends on the users' ability to process frequency and time information critical for speech perception. By identifying and enhancing this acoustic information, speech perception will significantly improve. In this AREA project, the investigators aim to establish and verify a tailored identification scheme for the spectral and temporal cues responsible for consonant recognition. The recent bimodal study conducted in the investigator's research laboratory shows that some frequency ranges and time segments of consonants are critical for consonant enhancement (called "target frequency or time ranges") while other frequency and time ranges cause consonant confusions (called "conflicting frequency or time ranges"). An Articulation Index-Gram (AI-Gram) signal processing can add and suppress intensity on these target and conflicting ranges. In Aim 1, the investigators will determine the effect of the dead regions on consonant recognition. Target and conflicting ranges will then be identified on an individual subject basis for each consonant in the HA alone, CI alone, and CI+HA in quiet. The target frequency range will be determined by finding the frequency regions creating dramatic consonant enhancement, while the conflicting frequency ranges will be determined by finding the frequency regions creating consonant confusion. The target time ranges will be determined by finding the segment of the consonants responsible for dramatic consonant improvement while systematically truncating the consonant. The target time range will be used as the conflicting time ranges because the conflicting frequency ranges would be the most detrimental factor affecting the target frequency ranges if they coincide in time. In Aim 2, consonant recognition will be measured in quiet and noise under the three AI-Gram processing conditions: 1) target ranges alone with +6 dB gain; 2) conflicting ranges alone with -6 dB suppression; and 3) both intensified target and suppressed conflicting ranges. For each AI-Gram processing condition, consonant recognition will be measured in the matched listening conditions (e.g., the target or conflicting ranges identified in the HA alone will be presented in the HA alone listening condition). To determine how the unilateral detection ability affects bimodal benefit, the consonants processed on the target or conflicting ranges identified in the HA alone and CI alone will each be presented to the CI+HA listening condition. This proposed work will identify acoustic cues that contribute to bimodal benefit and will reveal how these cues are integrated or interfered with across modalities. Defining the relative impact of the target and conflicting ranges on the AI-Gram-sensitive consonants in the HA alone, the CI alone, and the CI+HA together will help determine the upper and lower cutoff frequencies of a HA and a CI and fine-tune these cutoff frequencies. This data is much needed for the long-term goal: developing a tailored bimodal fitting procedure.

ELIGIBILITY:
Inclusion Criteria:

The proposed work requires the following qualifications to be met:

* be age from 18-74 years old,
* be native speakers of American English,
* be post-lingually deafened in both ears,
* be healthy enough to manipulate a computer mouse and read information on a computer monitor, and
* have at least 1-year of bimodal use prior to initiation of study participation to account for continuous improvement.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Bimodal benefit in percent correct scores for consonant perception with three signal processing conditions | 24 weeks
  Percent correct scores, ranging from minimum 0% to maximum 100% in consonant perception scores will be compared under three signal processing conditions: (1) when no signal processing is applied to consonants (baseline), (2) when the target frequency and time ranges responsible for consonant perception are intensified, and (3) when the conflicting frequency and time ranges causing consonant confusions are removed. Higher percent correct scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yang-Soo Yoon, PhD, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No